CLINICAL TRIAL: NCT06101693
Title: Biomarkers in Patients With Suspected Heart Failure With Preserved Ejection Fraction
Brief Title: Biomarkers in Patients With Suspected HFpEF
Acronym: BIOPEF
Status: Recruiting | Type: Observational
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other); Roche Diagnostics GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: GN23CA025
Record Dates: First submitted 2023-10-20; First posted 2023-10-26 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Heart Failure; Obesity; Heart Failure With Preserved Ejection Fraction
MeSH Terms: conditions — Heart Failure; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma RNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with NTproBNP<125ng/L and clinical suspicion of heart failure in primary care: Expected recruitment of 400 patients (50-60% expected prevalence of obesity, according to population study)
  Interventions: Diagnostic Test: Plasma biomarker levels
- Patients with NTproBNP125-399ng/L and clinical suspicion of heart failure in primary care: Expected recruitment of 400 patients (50% expected prevalence of obesity, according to population study)
  Interventions: Diagnostic Test: Plasma biomarker levels
- Patients with NTproBNP≥400ng/L and clinical suspicion of heart failure in primary care: Expected recruitment of 400 patients (50% expected prevalence of obesity, according to population study)
  Interventions: Diagnostic Test: Plasma biomarker levels

INTERVENTIONS:
Diagnostic Test: Plasma biomarker levels — This study will investigate the diagnostic utility and performance of:
  1. Alternative cut-offs for NT-proBNP to identify HF(pEF) in people with suspected HF and obesity, in whom
  2. Novel candidate biomarkers to identify HF(pEF) in people with suspected HF and obesity.
  3. Novel candidate biomarkers to identify HF(pEF) in people with suspected HF and NT-proBNP <125 ng/L
  4. The prevalence of HF in people with suspected HF and low NT-proBNP <125 ng/L).
  The diagnosis of heart failure will be determined according to international guidelines, when there are symptoms and/or signs of HF in association with "objective evidence of cardiac structural and/or functional abnormalities consistent with the presence of LV diastolic dysfunction/raised LV filling pressures". Non-invasive testing with rest and diastolic stress echocardiography will be used to evaluate for evidence of raised filling pressures, in order to make the study procedures applicable to usual clinical practice.
  Other Names: Rest echocardiography; Diastolic stress echocardiography

SUMMARY:
NT-proBNP does not adequately identify HF(pEF) in people with suspected HF at low levels, particularly in patients with obesity. This study will investigate:

1. alternative cut-offs for NT-proBNP to identify HF(pEF) in people with suspected HF and obesity
2. novel candidate biomarkers to identify HF(pEF) in people with suspected HF and obesity.
3. novel candidate biomarkers to identify HF(pEF) in people with suspected HF and NT-proBNP <125 ng/L
4. the prevalence of HF in people with suspected HF and low NT-proBNP <125 ng/L)

DETAILED DESCRIPTION:
This will be a prospective observational, non-randomised study of patients in primary care with suspected HF.

Detection of HFpEF in people without obesity is well-served by NT-proBNP. In contrast, NT-proBNP does not perform well when used to detect HFpEF in populations with obesity. There is increasing evidence that some people with low levels of NT-proBNP can have HF. As many as 50% of people with obesity and HFpEF (detected by elevated filling pressures) have NT-proBNP <125 ng/L. Some patients with HFpEF who are not obese can also have low natriuretic peptides levels.

Delayed diagnosis can lead to adverse outcomes for patients, in particular presentation acutely to secondary care. In addition to this, some patients with HFpEF who are not obese can also have low natriuretic peptides levels.

Patients with NTproBNP levels performed in the community for stable symptoms of suspected heart failure will be invited to participate.

Assessments in this study will include clinical history and examination, patient-reported outcome measures, electrocardiography, echocardiography and biomarker (blood and urine) analysis. Heart failure diagnostic scores and clinical evaluation by heart failure experts will be used to make a clinical diagnosis of heart failure, and to correlate this with levels of plasma and urine biomarkers, both established and novel.

Patients will be followed up passively (for a minimum of 10 years) using record linkage for subsequent hospitalisations or deaths.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age ≥ 18 years
* NT-proBNP sample taken by primary care physician as part of routine care for suspected heart failure

Exclusion Criteria:

* Unable to consent to inclusion in study due to significant cognitive impairment
* Geographical/ social reasons preventing attending study centre
* Unable to complete study assessments
* Patients presenting with acute HF or a previous diagnosis of HF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with NT-proBNP levels taken in primary care to evaluate for suspected heart failure will be invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 1028 (Estimated)
Dates: Start 2023-02-02 (Actual); Primary Completion 2025-09-29 (Estimated); Study Completion 2026-09-29 (Estimated)

PRIMARY OUTCOMES:
Optimal cut-offs for NT-proBNP to identify HFPEF in obese patients with suspected heart failure | 3 years
  To determine the utility and diagnostic performance of alternative cut-offs for NT-proBNP or combinations of biomarkers (including novel biomarker solutions)- with clinical variables to identify HFpEF in obese patients with suspected heart failure. (New biomarkers will be used for observational purposes only.)

SECONDARY OUTCOMES:
Prevalence of HF in patients with NT-proBNP<125ng/L | 3 years
  To identify the prevalence of HF in patients with NT-proBNP <125 ng/L with and without obesity, and suspected HF.
Optimal cut-offs for biomarkers to identify HFPEF in patients with suspected HF. | 3 years
  To determine the utility and diagnostic performance of alternative cut-offs for NT-proBNP or combinations of biomarkers (including novel biomarker solutions) with clinical variables to identify HFpEF in patients (with and without obesity) and suspected HF.
Utility and diagnostic performance of biomarkers (novel and adjusted stratified cut-offs) in patients with suspected HF (HFPEF, HFmREF, HFREF). | 3 years
  To determine the utility and diagnostic performance of novel biomarkers, adjusted N-terminal pro-B-type natriuretic peptide (NT-proBNP) cut-offs or combinations of biomarkers with clinical variables in patients with suspected HF (HFpEF, HFmrEF, HFrEF). (New biomarkers will be used for observational purposes only.)

CONTACTS AND LOCATIONS:
Overall Officials: Ross Campbell, MBChB, Principal Investigator — University of Glasgow
Locations (3):
- United Kingdom (3):
  - Glasgow Royal Infirmary, Glasgow
  - New Victoria Hospital, Glasgow
  - Queen Elizabeth University Hospital, Glasgow

REFERENCES:
- [Background] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J. 2021 Sep 21;42(36):3599-3726. doi: 10.1093/eurheartj/ehab368. No abstract available. PMID 34447992
- [Background] Madamanchi C, Alhosaini H, Sumida A, Runge MS. Obesity and natriuretic peptides, BNP and NT-proBNP: mechanisms and diagnostic implications for heart failure. Int J Cardiol. 2014 Oct 20;176(3):611-7. doi: 10.1016/j.ijcard.2014.08.007. Epub 2014 Aug 9. PMID 25156856
- [Background] Obokata M, Reddy YNV, Pislaru SV, Melenovsky V, Borlaug BA. Evidence Supporting the Existence of a Distinct Obese Phenotype of Heart Failure With Preserved Ejection Fraction. Circulation. 2017 Jul 4;136(1):6-19. doi: 10.1161/CIRCULATIONAHA.116.026807. Epub 2017 Apr 5. PMID 28381470
- [Background] Vaishnav J, Chasler JE, Lee YJ, Ndumele CE, Hu JR, Schulman SP, Russell SD, Sharma K. Highest Obesity Category Associated With Largest Decrease in N-Terminal Pro-B-Type Natriuretic Peptide in Patients Hospitalized With Heart Failure With Preserved Ejection Fraction. J Am Heart Assoc. 2020 Aug 4;9(15):e015738. doi: 10.1161/JAHA.119.015738. Epub 2020 Jul 30. PMID 32750299
- [Background] Buckley LF, Canada JM, Del Buono MG, Carbone S, Trankle CR, Billingsley H, Kadariya D, Arena R, Van Tassell BW, Abbate A. Low NT-proBNP levels in overweight and obese patients do not rule out a diagnosis of heart failure with preserved ejection fraction. ESC Heart Fail. 2018 Apr;5(2):372-378. doi: 10.1002/ehf2.12235. Epub 2018 Jan 18. PMID 29345112
- [Background] Meijers WC, Hoekstra T, Jaarsma T, van Veldhuisen DJ, de Boer RA. Patients with heart failure with preserved ejection fraction and low levels of natriuretic peptides. Neth Heart J. 2016 Apr;24(4):287-95. doi: 10.1007/s12471-016-0816-8. PMID 26940695
- [Background] Reddy YNV, Carter RE, Obokata M, Redfield MM, Borlaug BA. A Simple, Evidence-Based Approach to Help Guide Diagnosis of Heart Failure With Preserved Ejection Fraction. Circulation. 2018 Aug 28;138(9):861-870. doi: 10.1161/CIRCULATIONAHA.118.034646. PMID 29792299
- [Background] Pieske B, Tschope C, de Boer RA, Fraser AG, Anker SD, Donal E, Edelmann F, Fu M, Guazzi M, Lam CSP, Lancellotti P, Melenovsky V, Morris DA, Nagel E, Pieske-Kraigher E, Ponikowski P, Solomon SD, Vasan RS, Rutten FH, Voors AA, Ruschitzka F, Paulus WJ, Seferovic P, Filippatos G. How to diagnose heart failure with preserved ejection fraction: the HFA-PEFF diagnostic algorithm: a consensus recommendation from the Heart Failure Association (HFA) of the European Society of Cardiology (ESC). Eur J Heart Fail. 2020 Mar;22(3):391-412. doi: 10.1002/ejhf.1741. Epub 2020 Mar 5. PMID 32133741
- [Background] Sanders-van Wijk S, Barandiaran Aizpurua A, Brunner-La Rocca HP, Henkens MTHM, Weerts J, Knackstedt C, Uszko-Lencer N, Heymans S, van Empel V. The HFA-PEFF and H2 FPEF scores largely disagree in classifying patients with suspected heart failure with preserved ejection fraction. Eur J Heart Fail. 2021 May;23(5):838-840. doi: 10.1002/ejhf.2019. Epub 2020 Nov 2. No abstract available. PMID 33012125
- [Background] Popescu BA, Beladan CC, Nagueh SF, Smiseth OA. How to assess left ventricular filling pressures by echocardiography in clinical practice. Eur Heart J Cardiovasc Imaging. 2022 Aug 22;23(9):1127-1129. doi: 10.1093/ehjci/jeac123. No abstract available. PMID 35762650
- [Background] Guazzi M, Wilhelm M, Halle M, Van Craenenbroeck E, Kemps H, de Boer RA, Coats AJS, Lund L, Mancini D, Borlaug B, Filippatos G, Pieske B. Exercise testing in heart failure with preserved ejection fraction: an appraisal through diagnosis, pathophysiology and therapy - A clinical consensus statement of the Heart Failure Association and European Association of Preventive Cardiology of the European Society of Cardiology. Eur J Heart Fail. 2022 Aug;24(8):1327-1345. doi: 10.1002/ejhf.2601. Epub 2022 Jul 31. PMID 35775383
- [Background] Lancellotti P, Pellikka PA, Budts W, Chaudhry FA, Donal E, Dulgheru R, Edvardsen T, Garbi M, Ha JW, Kane GC, Kreeger J, Mertens L, Pibarot P, Picano E, Ryan T, Tsutsui JM, Varga A. The clinical use of stress echocardiography in non-ischaemic heart disease: recommendations from the European Association of Cardiovascular Imaging and the American Society of Echocardiography. Eur Heart J Cardiovasc Imaging. 2016 Nov;17(11):1191-1229. doi: 10.1093/ehjci/jew190. PMID 27880640
- [Background] Reddy YNV, Kaye DM, Handoko ML, van de Bovenkamp AA, Tedford RJ, Keck C, Andersen MJ, Sharma K, Trivedi RK, Carter RE, Obokata M, Verbrugge FH, Redfield MM, Borlaug BA. Diagnosis of Heart Failure With Preserved Ejection Fraction Among Patients With Unexplained Dyspnea. JAMA Cardiol. 2022 Sep 1;7(9):891-899. doi: 10.1001/jamacardio.2022.1916. PMID 35830183